CLINICAL TRIAL: NCT03227757
Title: Trial to Evaluate Treatment With Abbott Transcatheter Clip Repair System in Patients With Moderate or Greater Tricuspid Regurgitation (TRILUMINATE)
Brief Title: TRILUMINATE Study With Abbott Transcatheter Clip Repair System in Patients With Moderate or Greater TR
Acronym: TRILUMINATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-517
Record Dates: First submitted 2017-06-20; First posted 2017-07-24 (Actual); Results first posted 2021-10-26 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Tricuspid Valve Insufficiency
Keywords: TRILUMINATE; Percutaneous transcatheter intervention; Tricuspid regurgitation; Tricuspid Valve Repair System
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Tricuspid Valve Repair System (Experimental): Subjects who received TVRS will be included in this arm.
  Interventions: Device: Tricuspid Valve Repair System

INTERVENTIONS:
Device: Tricuspid Valve Repair System — Subjects who received TVRS will be included in this arm. The TVRS is intended for reconstruction of the insufficient tricuspid valve through tissue approximation.

SUMMARY:
The primary purpose of this study is to evaluate safety and effectiveness of the Tricuspid Valve Repair System (TVRS) for treating symptomatic moderate or greater tricuspid regurgitation (TR) in patients currently on medical management and who are deemed appropriate for percutaneous transcatheter intervention.

DETAILED DESCRIPTION:
This is a prospective, single arm, multi-center study.

A minimum of 85 subjects will be prospectively enrolled into this single arm study in approximately 25 sites, in Europe, Canada and the United States. Patients will be seen for follow-up visits at discharge (≤ 7 days post index procedure), 30 days, 6 months, 1,2,3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥18 years and ≤ 90 years at time of consent and must not be a member of a vulnerable population.
2. Subject or a legally authorized representative (where allowed per local regulations) must provide written informed consent prior to any trial related procedure.
3. Subject must agree not to participate in any other clinical trial for a period of one year following the index procedure.
4. In the judgment of the investigator at the site, the subject has been adequately treated per applicable standards, including for coronary artery disease, mitral regurgitation and heart failure at least 30-days prior to index procedure. The Eligibility Committee must concur that the subject has been adequately treated.
5. New York Heart Association (NYHA) Functional Class II (conditional), III, or ambulatory IV

   1. Subjects with moderate TR: Only NYHA Class III or IV may be considered
   2. Subjects with severe or greater TR: NYHA II, III, or IV may be considered for inclusion
6. No indication for left-sided or pulmonary valve correction.
7. The Site Heart Team concur the benefit-risk analysis supports intervention for tricuspid regurgitation per current guidelines for the management of Valvular heart disease and that the subject is at high risk for tricuspid valve surgery.
8. In the judgement of the TVRS implanting investigator, femoral vein access is determined to be feasible and can accommodate a 25 Fr catheter.

   Echocardiographic Inclusion Criteria:
9. Moderate or greater (≥2+) Tricuspid Regurgitation determined by the assessment of a qualifying transthoracic echocardiogram (TTE) and transesophageal echocardiogram (TEE) confirmed by the Echocardiography Core Lab (ECL).
10. Tricuspid valve anatomy determined to be suitable for implantation determined by the site heart team.
11. Tricuspid valve anatomy evaluable by TTE and TEE.

Exclusion Criteria:

1. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.
2. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.
3. Severe uncontrolled hypertension (Systolic blood pressure [SBP] ≥ 180 mmHg and/or Diastolic blood pressure [DBP] ≥ 110 mm Hg).
4. Systolic Pulmonary Artery Pressure > 60 mmHg (echo determined).
5. Prior tricuspid valve leaflet surgery or any currently implanted prosthetic tricuspid valve, or any prior transcatheter tricuspid valve procedure.
6. Mitral Regurgitation moderate-severe or greater severity (≥3+).
7. Pacemaker or implantable cardioverter-defibrillator (ICD) leads that would prevent appropriate placement of TVRS Clip.
8. Active endocarditis or active rheumatic heart disease or leaflets degenerated from rheumatic disease.
9. Myocardial Infarction (MI) or known unstable angina within prior 30 days prior to enrollment.
10. Percutaneous coronary intervention within prior 30 days prior to enrollment.
11. Hemodynamic instability defined as systolic pressure < 90 mmHg with or without afterload reduction, cardiogenic shock or the need for inotropic support or intra-aortic balloon pump or other hemodynamic support device.
12. Cerebrovascular Accident (CVA) within prior 3 months to enrollment.
13. Chronic dialysis.
14. Bleeding disorders or hypercoagulable state.
15. Active peptic ulcer or active gastrointestinal (GI) bleeding.
16. Contraindication, allergy or hypersensitivity to dual antiplatelet and anticoagulant therapy.
17. Active infections requiring current antibiotic therapy (if temporary illness, patients may enroll 4 weeks after discontinuation of antibiotics with no active infection).
18. Known allergy or hypersensitivity to device materials.
19. In the judgement of the investigator, a condition that could limit a patient's ability or unwillingness to participate in the study, comply with study required testing and/or follow-up visits or that could impact scientific integrity of the study.
20. Evidence of intracardiac, inferior vena cava (IVC), or femoral venous mass, thrombus or vegetation.
21. Life expectancy of less than 12 months due to non-cardiac conditions.

    Echocardiographic Exclusion Criteria:
22. Tricuspid stenosis.
23. Left Ventricular Ejection Fraction (LVEF) ≤20%.
24. Tricuspid valve leaflet anatomy which may preclude clip implantation, proper clip positioning on the leaflets or sufficient reduction in TR. This may include:

    1. Evidence of calcification in the grasping area
    2. Presence of a severe coaptation defect (> 2cm) of the tricuspid leaflets

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Georg Nickenig, Principal Investigator — University Hospital, Bonn
Locations (20):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Henry Ford Hospital, Detroit, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mount Sinai Hospital, New York, New York
- France (2):
  - Hospital Nord Laennec - Chu De Nantes, Nantes, Saint-Herblain
  - Bichat-Claude Bernard Hospital, Paris
- Germany (6):
  - Ludwig-Maximilian University of Munich (LMU), Munich, Bavaria
  - Schuchtermann Klinik, Bad Rothenfelde, Lower Saxony
  - University Hospital Bonn, Bonn, North Rhine-Westphalia
  - Universitatsmedizin der Johannes Gutenberg-Universitat Mainz, Mainz, Rhineland-Palatinate
  - Leipzig Heart Center, Leipzig, Saxony
  - Albertinen-Krankenhaus, Hamburg
- Italy (3):
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele - Presidio Ferrarotto, Catania, Catania (CT)
  - San Raffaele University Hospital, Milan, Milan
  - Istituto Clinico Sant'Ambrogio, Milan, Milan
- Spain (2):
  - Hospital de Sant Pau, Barcelona
  - Clinical and Provincial Hospital of Barcelona, Barcelona
- Switzerland (3):
  - Inselspital Bern, Bern
  - HerzKlinik Hirslanden - Klinik Hirslanden, Zurich
  - University Hospital of Zurich (USZ), Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nickenig G, Lurz P, Sorajja P, von Bardeleben RS, Sitges M, Tang GHL, Hausleiter J, Trochu JN, Nabauer M, Heitkemper M, Ying SW, Weber M, Hahn RT; TRILUMINATE Investigators. Percutaneous Edge-to-Edge Repair for Tricuspid Regurgitation: 3-Year Outcomes From the TRILUMINATE Study. JACC Cardiovasc Interv. 2024 Sep 23;17(18):2113-2122. doi: 10.1016/j.jcin.2024.05.036. Epub 2024 Sep 4. PMID 39243264
- [Derived] von Bardeleben RS, Lurz P, Sorajja P, Ruf T, Hausleiter J, Sitges M, Da Rocha E Silva J, Nabauer M, Weber M, Tang GHL, Heitkemper M, Ying SW, Trochu JN, Kar S, Hahn RT, Nickenig G; TRILUMINATE Trial Investigators. Two-Year Outcomes for Tricuspid Repair With a Transcatheter Edge-to-Edge Valve Repair From the Transatlantic TRILUMINATE Trial. Circ Cardiovasc Interv. 2023 Aug;16(8):e012888. doi: 10.1161/CIRCINTERVENTIONS.122.012888. Epub 2023 Aug 15. PMID 37582170
- [Derived] Lurz P, Stephan von Bardeleben R, Weber M, Sitges M, Sorajja P, Hausleiter J, Denti P, Trochu JN, Nabauer M, Tang GHL, Biaggi P, Ying SW, Trusty PM, Dahou A, Hahn RT, Nickenig G; TRILUMINATE Investigators. Transcatheter Edge-to-Edge Repair for Treatment of Tricuspid Regurgitation. J Am Coll Cardiol. 2021 Jan 26;77(3):229-239. doi: 10.1016/j.jacc.2020.11.038. PMID 33478646
- [Derived] Nickenig G, Weber M, Lurz P, von Bardeleben RS, Sitges M, Sorajja P, Hausleiter J, Denti P, Trochu JN, Nabauer M, Dahou A, Hahn RT. Transcatheter edge-to-edge repair for reduction of tricuspid regurgitation: 6-month outcomes of the TRILUMINATE single-arm study. Lancet. 2019 Nov 30;394(10213):2002-2011. doi: 10.1016/S0140-6736(19)32600-5. Epub 2019 Nov 7. PMID 31708188

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 98 subjects were enrolled and underwent Tricuspid Valve Repair System (TVRS) procedure.
Period: Overall Study
Arm/Group | Tricuspid Valve Repair System
Started | 98
Completed | 60
Not Completed | 38
Not completed — Death | 25
Not completed — Withdrawal | 10
Not completed — Missed visits | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tricuspid Valve Repair System
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The number of participants analyzed includes subjects who were available at that time of analysis
  Participants
    Ethnicity: number analyzed (Participants) | 71
    Ethnicity: Hispanic or Latino | 6
    Ethnicity: Unknown or Not Reported | 65
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
  France | 2
  Germany | 45
  Italy | 11
  Spain | 8
  Switzerland | 7
New York Heart Association (NYHA) class II or above [Count of Participants; unit: Participants] — NYHA functional classification system relates symptoms to everyday activities and the patient's quality of life.
  NYHA Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  NYHA Class II: Subjects with cardiac disease resulting in slight limitation of physical activity.
  NYHA Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  NYHA Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort. Population: The number of participants analyzed includes subjects who were available at that time of analysis
  Participants
    number analyzed (Participants) | 96
    NYHA class I | 0
    NYHA class II | 23
    NYHA class III | 69
    NYHA class IV | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Echocardiographic Tricuspid Regurgitation Reduction at Least 1 Grade
Description: Tricuspid regurgitation (TR) was assessed with standard 2D color doppler methods using a integrative approach. A five-class grading scheme was used: mild, moderate, severe, massive and torrential. Parameters including vena contracta area, effective regurgitant orifice area and proximal isovelocity surface area were used to quantify and grade TR.
Time Frame: At 30 days
Population: The first 85 enrolled subjects with an attempted TriClip™ procedure upon femoral vein puncture. Note: The sample size and power estimation specified in the clinical investigation protocol indicated that a total of 85 subjects provided sufficient power to evaluate the primary endpoints. This endpoint was assessed in 82 of the 85 subjects. The reason for the inability to assess the endpoint in 3 subjects was missing echocardiogram data and limited imaging quality at baseline (1) and 30 days (2).
Measure: Count of Participants; unit: Participants
Arm/Group | Tricuspid Valve Repair System
Number analyzed (Participants) | 82
Participants | 71

2. Primary Outcome: Number of Participants With Composite of Major Adverse Event (MAE)
Description: Major Adverse Event (MAE) is defined as a composite of:
  * Cardiovascular Mortality
  * Myocardial Infarction (MI)
  * Stroke
  * New onset renal failure
  * Endocarditis requiring surgery, and
  * Non-elective cardio-vascular (CV) surgery for TVRS device-related AE post-procedure
Time Frame: At 6 months
Population: The first 85 enrolled subjects with an attempted TriClip™ procedure upon femoral vein puncture. Note: The sample size and power estimation specified in the clinical investigation protocol indicated that a total of 85 subjects provided sufficient power to evaluate the primary endpoints. One subject withdrew from the study prior to the early window of the 6-month visit, without any reported adverse events, and was therefore excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Tricuspid Valve Repair System
Number analyzed (Participants) | 84
Participants | 5

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Tricuspid Valve Repair System
All-Cause Mortality (participants affected / at risk) | 25/98
Serious Adverse Events (participants affected / at risk) | 68/98
Other Adverse Events (participants affected / at risk) | 88/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tricuspid Valve Repair System (N=98)
ANAEMIA (Blood and lymphatic system disorders) | 2
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1
HAEMORRHAGIC DIATHESIS (Blood and lymphatic system disorders) | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 5
Atrial flutter (Cardiac disorders) | 5
CARDIAC ARREST (Cardiac disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 21
Cardiorenal syndrome (Cardiac disorders) | 3
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 2
Sick sinus syndrome (Cardiac disorders) | 1
TACHYARRHYTHMIA (Cardiac disorders) | 1
Tricuspid valve incompetence (Cardiac disorders) | 3
Vertigo (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 1
PANCREATITIS (Gastrointestinal disorders) | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 1
ASTHENIA (General disorders) | 1
Chest pain (General disorders) | 2
DEVICE DEPLOYMENT ISSUE (General disorders) | 1
DEVICE MALFUNCTION (General disorders) | 2
Death (General disorders) | 3
Multi-organ failure (General disorders) | 2
POLYP (General disorders) | 1
SUDDEN DEATH (General disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
CORONA VIRUS INFECTION (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
Gallbladder empyema (Infections and infestations) | 1
INFECTION (Infections and infestations) | 2
PNEUMONIA VIRAL (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 8
SEPSIS (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 1
BURNS SECOND DEGREE (Injury, poisoning and procedural complications) | 1
CONTUSION (Injury, poisoning and procedural complications) | 1
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1
FALL (Injury, poisoning and procedural complications) | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Blood sodium decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
FLUID RETENTION (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BREAST CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MYELOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2
EPILEPSY (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
VIITH NERVE PARALYSIS (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 12
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
ARRHYTHMIA PROPHYLAXIS (Surgical and medical procedures) | 1
Arteriovenous fistula (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Femoral arterial stenosis (Vascular disorders) | 1
HAEMATOMA (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 19
Hypertension (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
VENOUS INSUFFICIENCY (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tricuspid Valve Repair System (N=98)
ANAEMIA (Blood and lymphatic system disorders) | 3
ANAEMIA MACROCYTIC (Blood and lymphatic system disorders) | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1
HAEMORRHAGIC DIATHESIS (Blood and lymphatic system disorders) | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1
ANGINA PECTORIS (Cardiac disorders) | 2
ATRIAL FLUTTER (Cardiac disorders) | 5
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 8
BRADYCARDIA (Cardiac disorders) | 4
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 1
CARDIAC ARREST (Cardiac disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
CARDIORENAL SYNDROME (Cardiac disorders) | 3
CHORDAE TENDINAE RUPTURE (Cardiac disorders) | 2
CORONARY ARTERY DISEASE (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 28
INTRACARDIAC THROMBUS (Cardiac disorders) | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 4
MYOCARDIAL INFARCTION (Cardiac disorders) | 3
PERICARDIAL EFFUSION (Cardiac disorders) | 2
SICK SINUS SYNDROME (Cardiac disorders) | 1
TACHYARRHYTHMIA (Cardiac disorders) | 1
TACHYCARDIA (Cardiac disorders) | 2
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 8
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 1
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 2
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 1
HYPERTHYROIDISM (Endocrine disorders) | 1
CATARACT (Eye disorders) | 1
GLAUCOMA (Eye disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 2
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1
OESOPHAGITIS ULCERATIVE (Gastrointestinal disorders) | 1
PANCREATITIS (Gastrointestinal disorders) | 1
TOOTH DISORDER (Gastrointestinal disorders) | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 1
ASTHENIA (General disorders) | 1
CATHETER SITE HAEMATOMA (General disorders) | 1
CHEST PAIN (General disorders) | 6
DEATH (General disorders) | 3
DEVICE DEPLOYMENT ISSUE (General disorders) | 4
DEVICE MALFUNCTION (General disorders) | 2
FATIGUE (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1
IMPAIRED HEALING (General disorders) | 1
MULTI-ORGAN FAILURE (General disorders) | 2
OEDEMA (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 2
PAIN (General disorders) | 2
POLYP (General disorders) | 2
PYREXIA (General disorders) | 1
SUDDEN DEATH (General disorders) | 1
THROMBOSIS IN DEVICE (General disorders) | 1
CHOLESTASIS (Hepatobiliary disorders) | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 1
LIVER INJURY (Hepatobiliary disorders) | 1
SEASONAL ALLERGY (Immune system disorders) | 1
BACTERIAL INFECTION (Infections and infestations) | 1
BRONCHITIS (Infections and infestations) | 1
BRONCHOPNEUMONIA (Infections and infestations) | 1
CANDIDIASIS (Infections and infestations) | 1
CORNEAL INFECTION (Infections and infestations) | 1
CORONA VIRUS INFECTION (Infections and infestations) | 1
ERYSIPELAS (Infections and infestations) | 1
GALLBLADDER EMPYEMA (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
HERPES ZOSTER (Infections and infestations) | 1
INFECTION (Infections and infestations) | 5
INFLUENZA (Infections and infestations) | 2
PHARYNGITIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 8
PNEUMONIA VIRAL (Infections and infestations) | 2
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
RHINITIS (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 3
UROSEPSIS (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 8
ARTHROPOD STING (Injury, poisoning and procedural complications) | 1
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 1
BURNS SECOND DEGREE (Injury, poisoning and procedural complications) | 1
CONTUSION (Injury, poisoning and procedural complications) | 1
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1
FALL (Injury, poisoning and procedural complications) | 8
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 1
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 1
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1
ANTICOAGULATION DRUG LEVEL BELOW THERAPEUTIC (Investigations) | 1
BLOOD CREATININE INCREASED (Investigations) | 1
BLOOD PRESSURE INCREASED (Investigations) | 1
BLOOD SODIUM DECREASED (Investigations) | 1
CARDIOACTIVE DRUG LEVEL DECREASED (Investigations) | 2
COAGULATION FACTOR DECREASED (Investigations) | 1
HAEMOGLOBIN DECREASED (Investigations) | 2
HEART RATE INCREASED (Investigations) | 1
N-TERMINAL PROHORMONE BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 1
OCCULT BLOOD (Investigations) | 1
OXYGEN SATURATION DECREASED (Investigations) | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 2
FLUID RETENTION (Metabolism and nutrition disorders) | 1
GOUT (Metabolism and nutrition disorders) | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 4
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 1
ADRENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BREAST CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MYELOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
ANOSMIA (Nervous system disorders) | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2
CONVULSION (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 2
EPILEPSY (Nervous system disorders) | 1
MYOCLONUS (Nervous system disorders) | 1
PARAESTHESIA (Nervous system disorders) | 2
POLYNEUROPATHY (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 3
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1
VIITH NERVE PARALYSIS (Nervous system disorders) | 1
VOCAL CORD PARALYSIS (Nervous system disorders) | 1
ANXIETY (Psychiatric disorders) | 1
ANXIETY DISORDER DUE TO A GENERAL MEDICAL CONDITION (Psychiatric disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1
DELIRIUM (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 1
INSOMNIA (Psychiatric disorders) | 1
MENTAL DISORDER DUE TO A GENERAL MEDICAL CONDITION (Psychiatric disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 21
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2
URINARY RETENTION (Renal and urinary disorders) | 1
BREAST PAIN (Reproductive system and breast disorders) | 1
GYNAECOMASTIA (Reproductive system and breast disorders) | 2
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 10
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1
HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2
DERMAL CYST (Skin and subcutaneous tissue disorders) | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 1
ARRHYTHMIA PROPHYLAXIS (Surgical and medical procedures) | 1
STOMACH DILATION PROCEDURE (Surgical and medical procedures) | 1
ARTERIOVENOUS FISTULA (Vascular disorders) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 3
EMBOLISM (Vascular disorders) | 1
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 1
HAEMATOMA (Vascular disorders) | 3
HYPERTENSION (Vascular disorders) | 3
HYPERTENSIVE CRISIS (Vascular disorders) | 2
HYPOTENSION (Vascular disorders) | 5
Haemorrhage (Vascular disorders) | 31
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1
VENOUS INSUFFICIENCY (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT03227757/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT03227757/SAP_001.pdf